CLINICAL TRIAL: NCT07337616
Title: Clinical Assessment of Field Shield Wound Dressing of Large Surface Area Burn Wounds
Brief Title: Field Shield Wound Dressing Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: KeriCure Medical (Industry)
Collaborators: Valleywise Health (Other); United States Army Institute of Surgical Research (U.S. Federal Agency); The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20240572
Record Dates: First submitted 2026-01-08; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Burn Wounds - Partial Thickness (2nd Degree)
Keywords: FSWD; Burn wounds
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: In this study each subject will serve as their own control receiving the intervention dressing on one wound and the standard of care dressing on another wound.
Who Masked: Participant, Outcomes Assessor
Masking Description: Only the individual performing dressing changes will know which dressing is applied to which site. All others will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- FSWD wound site (Experimental): One burn wound site on each participant will receive study treatment.
  Interventions: Device: Field Shield Wound Dressing
- Control treatment (Active Comparator): One burn wound site on each patient receives standard treatment with silver dressing.
  Interventions: Device: Silverlon

INTERVENTIONS:
Device: Field Shield Wound Dressing — Spray on wound dressing.
  Arms: FSWD wound site
Device: Silverlon — Silver dressing
  Arms: Control treatment

SUMMARY:
This study is to compare the Field Shield Wound Dressing (FSWD) as a treatment for burn wounds to a standard of care burn wound dressing to evaluate healing, infection, pain/discomfort, and deepening of wound over time.

DETAILED DESCRIPTION:
To assess FSWD in comparison to standard of care dressing, subjects will undergo dressing changes and visual assessments.

ELIGIBILITY:
Inclusion Criteria:

* Thermal injury size 5-30% TBSA
* Admitted to the burn center and enroll able within 72 hours of injury
* Subject has two distinct areas of 100cm2 or larger of intermediate to deep partial thickness burns (study sites). These areas are judged to be comparable in depth.
* The subject and or caregiver is able and willing to follow the protocol requirements
* Achieve wound photos and dressing change at 3 days

Exclusion Criteria:

* Subject has congestive heart failure, oxygen-dependent chronic lung disease, end-stage renal disease, or liver cirrhosis

  * Subject is undergoing hospice care.
  * Subject is currently being treated for an active malignant disease
  * Subject has other concurrent conditions that in the opinion of the Investigator may compromise subject safety
  * Known contraindications to silver metals, silver chloride, or silver tetraoxide
  * Known contraindications to lidocaine
  * Known allergies to any components of either primary dressing in the study
  * Known allergies to the silicone or adhesives in secondary dressings
  * Burns located on the hands, feet, face, and/or genitals will be excluded from treatment sites, but will be included in the total TBSA calculation
  * Subject has a combined TBSA of 31% or greater of partial and/or full thickness burn wounds
  * Concurrent participation in another clinical trial that involves an investigational drug or device that would interfere with this study.
  * Subject is pregnant, breast feeding, or planning to become pregnant.
  * Subjects who, within 60 days prior to enrollment, have a history of more than two weeks treatment with immunosuppressants (including systemic corticosteroids >10mg daily dose), cytotoxic chemotherapy, application of topical steroids within one month prior to enrollment, or who receive such medications during the screening period, or who are anticipated to require such medications during the course of the study.
  * Burn study site(s) has been previously treated with tissue engineered materials (e.g., Apligraf® or Dermagraft®) or other scaffold materials (e.g., Oasis, Matristem) preceding the study wound dressing application.
  * Burn study site(s) has been previously treated with a silvadene

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-09-29 (Estimated)

PRIMARY OUTCOMES:
Wound closure | From enrollment to end of study, 4-6 months.
  Wound closure will be assessed at each time point (day 3, 7, 12, 19, 28, 35). The probability of wound closure will be assessed with a cluster randomized Generalized Estimating Equations (GEE) model of the probability of closure in terms of treatment and clinical site with clustering by patient and login link.

SECONDARY OUTCOMES:
Infection | 35 days
  Rate of occurrence of infection per uint time.
Surgical debridement | 35 days
  Rate of occurrence of surgical debridement and rate of occurrence of grafting
Pain severity | days 3, 7, 12, 19, and 28.
  Pain will measured using a visual analog scale (0-10) at each dressing change comparing each site pain ratings.
Scar | day 35 and 4-6 months
  The Patient and Observer Scar Assessment Scale will be conducted to evaluate scars, comparing the two sites at two time points.
Health-related quality of life | day 35 and 4-6 months
  A burn specific health-related quality of life assessment will be conducted and compared at two time points.
Function | Day 3, 35 and 4-6 months
  The Patient Specific Function Scale assessment will be conducted and compared at three time points

CONTACTS AND LOCATIONS:
Overall Officials: Kerriann Greenhalgh, PH.D., Principal Investigator — KeriCure Medical
Locations (2):
- United States (2):
  - Valleywise Health, Phoenix, Arizona
  - United State Army Institute of Surgical Research, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
All collected de-identified IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: January 1, 2027
Access Criteria: Data will be submitted to the National Trauma Research Repository. Access will be limited to investigators with approved access.